CLINICAL TRIAL: NCT03233815
Title: Benefits of Total Intravenous Anesthesia Compared With Inhaled Anesthesia in Cardiovascular Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2017-3604-95
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Surgical Procedure
Keywords: Inhaled anesthesia; Total intravenous anesthesia
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inhaled anesthesia (Sevoflurane): Patients undergoing cardiovascular surgery with inhaled anesthesia with sevoflurane.
  Interventions: Drug: Sevoflurane
- Total Intravenous Anesthesia (Propofol): Patients undergoing cardiovascular surgery with total intravenous anesthesia with propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol anesthesia Dose: 4-6mg/kg/h
  Other Names: Diprivan
  Groups: Total Intravenous Anesthesia (Propofol)
Drug: Sevoflurane — Inhaled anesthesia with sevoflurane. Dose: 1-2.5 Minimum Alveolar Concentration(MAC)
  Other Names: Sevorane
  Groups: Inhaled anesthesia (Sevoflurane)

SUMMARY:
This study compares the difference in proinflammatory markers Interleukin 6 (IL-6), Tumor necrosis factor alpha (TNFα) and cortisol in patients undergoing cardiovascular surgery to asses if there is a benefit of using intravenous total anesthesia (TIVA) over inhaled anesthesia for this procedures.

DETAILED DESCRIPTION:
IL-6, TNFα and cortisol will be measure at the beginning of the cardiovascular surgery and 20 minutes after the cardiovascular bypass ends to calculate the difference between them and compare if there is any statistical difference between the proinflammatory markers with the two anesthesia techniques.

ELIGIBILITY:
Inclusion Criteria:

Scheduled for cardiovascular surgery American Society of Anaesthesiologists (ASA) physical status classification II-IV BMI < 25 HbA1c < 7%

Exclusion Criteria:

Diabetic patients Known allergy to propofol

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for cardiovascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-11-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
IL-6 | The difference between IL-6 at the begging of surgery and 20 minutes after the end of the cardiopulmonary bypass
  IL-6 will be compared between the groups.

SECONDARY OUTCOMES:
TNFα | The difference between TNFα at the begging of surgery and 20 minutes after the end of the cardiopulmonary bypass
  TNFα will be compared between the groups
Cortisol | The difference between cortisol at the begging of surgery and 20 minutes after the end of the cardiopulmonary bypass
  Cortisol will be compared between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gallardo, PhD, Principal Investigator — Instituto Mexicano del Seguroa Social
Locations (1):
- Hospital de cardiología, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The plan is not decided yet.